CLINICAL TRIAL: NCT06649318
Title: Effect of Brain GABA Metabolite Amount to Propofol Utilisation Under TIVA in Hypothyroid Patient
Acronym: BrainGABA
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-117
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hypothyroidism; Anesthesia, General; Propofol Dosage; Magnetic Resonance Imaging (MRI); Remifentanil; Gamma Aminobutyric Acid
Keywords: Hypothyroid patient; GABA metabolites; Magnetic resonance spectroscopy screening; propofol; remifentanyl; anesthesia
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Control group (n=40) Patients with normal thyroid function tests
- Group 2: Hypothyroid patients group (n=40) . Hypothyroid and treated with Levothyroxine

SUMMARY:
Introduction: GABAergic synaptic transmigration in the anterior cingulate (ACC) cortex of hypothyroid rats has been demonstrated by electrophysiologic recordings. In this study, the investigators primary aim was to determine whether the dose requirement of propofol used under the guidance of bispectral index monitoring is correlated with thyroid hormone levels in patients undergoing surgery under total intravenous anaesthesia.The investigators secondary aim was to determine whether there is a difference in the amount of GABA metabolite in the midline posterior (mPCC) and midline anterior cingulate cortex (mACC) region in normal and thyroid dysfunction patients on magnetic resonance spectroscopic imaging.

Method: After ethics committee approval, the study included patients with ASA I-II status: Group 1 (Control group n=40) patients with regular thyroid function tests and Group 2 (Hypothyroid group n=40) patients with hypothyroidism history with Levothyroxine sodium treated. Patients were evaluated preoperatively with the Montreal assessment scale and Beck anxiety scale. Written informed consent was obtained from all the patients, andparticipants underwent a brain MRI examination one day before the operation. The possible increase of GABA, which is present in the imaging with NAA, Cr and Glx in the range of 2.2-2.4 ppm, was recorded as an elevated spectral curve in the MR spectroscopy spectrum and its numerical equivalent was determined as the amount of chemical shifting in the y-axis. To determine GABA, the investigators set the sequence with optimal parameters, for which the investigators set the radio frequency pulse-echo time (TE) as 20 msec.The investigators set the voxel size as 2*3*3 cm to obtain optimal results. Researchers determined single voxel imaging MR spectroscopy sampling area in the midline anterior and posterior to the cingulate gyrus in all patients. Patients with spectral voxels outside the specified area, dense ventricular contamination within the voxel, or with intra-voxel dense ventricular contamination or seminal contamination were excluded from the study.

Patients were operated on under total intravenous anaesthesia. Anesthesia Induction was performed with 2 mg/kg propofol, 0.5 mg/kg fentanyl and 0.5 mg/kg rocuronium. Maintenance was achieved by bispectral index monitoring with propofol infusion at a dose of 1-8 mg/kg/min and remifentanil infusion at a dose of 0.5-2 mcg/kg/min with values between 40-60.

DETAILED DESCRIPTION:
It is generally accepted that thyroid hormones have important effects on the normal functioning of the adult brain. Hypothyroidism is a common endocrine disorder characterized by low secretion of thyroid hormone. It is often associated with cognitive and neuropsychiatric changes. Multimodal imaging studies have demonstrated structural and functional changes in the brain in patients with hypothyroidism. Publications have reported decreased hippocampal area, microstructural changes in brain white matter, changes in brain metabolic rate, decreased regional blood flow, decreased cerebral glucose metabolism, decreased functional connectivity and decreased cortical excitability.

It is noteworthy that the hormone affects GABAergic neurotransmission. Preclinical studies have shown that T3 and T4 hormones modulate GABA receptor activity. Recent studies in rat hippocampus have shown a decrease in GABA levels in the hippocampus in the hypothyroid group. Anesthetic drugs that researchers use as daily routine anesthetic applications in the clinic for general anesthesia mostly show their effects through GABA receptors. Therefore, the investigators argue that in thyroid hormone disorders, which are effective on the GABAergic system, the need for anesthetic substances routinely used during general anesthesia may vary compared to patients with normal thyroid function.

The investigators study, they aimed to observe whether there is a difference between the anesthetic substance requirements of patients with normal thyroid function and hypothyroid patients under general anesthesia with monitoring. The researchers also aimed to observe whether there is a regional difference in non-contrast MR spectroscopic evaluation in patients with normal and low thyroid dysfunction. There were no invasive procedures in the investigators study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and younger than 65 years who will be operated under total intravenous anesthesia
* ASAI-II status

Exclusion Criteria:

* Patients for whom Intensive Care Unit (ICU) indication is foreseen
* Chronic obstructive pulmonary disease,
* A personal or family history of malignant hyperthermia,
* Alcohol or drug addiction,
* History of liver or kidney disease,
* With coronary artery disease or heart failure,
* Significant anemia or hemoglobinopathy,
* Hypotension, hypovolemia, sepsis,
* Unregulated diabetic patients,
* Female patients who are pregnant or lactating.
* Allergic to propofol and halogens
* Patients on gabapentinoids
* Those with a history of head trauma
* Those with neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients ASAI-II status, older than 18 years and younger than 65 years who will be operated under total intravenous anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Changes of participants' thyroid hormone levels measured before anesthesia and doses of propofol and remifentanil used in total intravenous anesthesia under bispectral index monitoring. | From enrollment to the end of treatment at 1 day
  The difference of participants' thyroid hormone levels (IU/mL) before anesthesia and compare the doses of propofol in miligram and remifentanil in microgram used in total intravenous anesthesia under bispectral index monitoring.

SECONDARY OUTCOMES:
Changes in the amounts of brain GABA metabolites chemical shifts measured in ppm units between participants with hypothyroidism and participants with normal thyroid function before anesthesia. . | From enrollment to the end of treatment at 1 day
  To determine whether there is a difference in the amount of GABA metabolite in the midline posterior (mPCC) and midline anterior cingulate cortex (mACC) region in normal and thyroid dysfunction patients on magnetic resonance spectroscopic imaging and its correlation of the propofol and remifentanil needing.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, DU, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brohan J, Goudra BG. The Role of GABA Receptor Agonists in Anesthesia and Sedation. CNS Drugs. 2017 Oct;31(10):845-856. doi: 10.1007/s40263-017-0463-7. PMID 29039138
- [Background] Fu X, Sun P, Zhang X, Zhu D, Qin Q, Lu J, Wang J. GABA in the anterior cingulate cortex mediates the association of white matter hyperintensities with executive function: a magnetic resonance spectroscopy study. Aging (Albany NY). 2024 Mar 1;16(5):4282-4298. doi: 10.18632/aging.205585. Epub 2024 Mar 1. PMID 38441529
- [Background] Yi J, Zheng JY, Zhang W, Wang S, Yang ZF, Dou KF. Decreased pain threshold and enhanced synaptic transmission in the anterior cingulate cortex of experimental hypothyroidism mice. Mol Pain. 2014 Jun 18;10:38. doi: 10.1186/1744-8069-10-38. PMID 24943008